CLINICAL TRIAL: NCT06922604
Title: A Phase 1b Study of Glofitamab in CNS Lymphoma
Brief Title: Glofitamab With Obinutuzumab Pre-treatment for the Treatment of Central Nervous System Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24487; NCI-2025-02019 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24487 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Primary Central Nervous System Lymphoma; Secondary Central Nervous System Lymphoma
MeSH Terms: interventions — Specimen Handling; glofitamab; Spinal Puncture; Magnetic Resonance Spectroscopy; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (obinutuzumab, glofitamab) (Experimental): Patients receive obinutuzumab IV on day 1 of cycle 1 and glofitamab IV over 2-4 hours on days 8 and 15 of cycle 1 and on day 1 of subsequent cycles. Cycles repeat every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo CT or PET/CT at screening and CSF and blood sample collection, brain MRI throughout the study. Patients with secondary CNS lymphoma also undergo CT or PET/CT throughout the study. Additionally, patients with baseline CSF involvement, may undergo lumbar puncture throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Glofitamab; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Biological: Obinutuzumab; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo CSF and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT or PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Glofitamab — Given IV
  Other Names: Anti-CD20 x Anti-CD3 Bispecific Monoclonal Antibody RO7082859; Columvi; Glofitamab-gxbm; RO 7082859; RO-7082859; RO7082859
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Magnetic Resonance Imaging — Undergo brain MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA 101; GA-101; GA101; Gazyva; huMAB(CD20); R 7159; R-7159; R7159; RO 5072759; RO-5072759; RO5072759
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This phase Ib trial tests the safety and side effects of glofitamab after pre-treatment with obinutuzumab and how well they work in treating patients with central nervous system (CNS) lymphoma. Glofitamab is a bispecific antibody that can bind to two different antigens (substances that cause the body to make a specific immune response) at the same time. Glofitamab binds to CD20 on lymphoma cells, and CD3 on T-cells (a type of white blood cell) and may interfere with the ability of cancer cells to grow and spread. Obinutuzumab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Obinutuzumab can also be administered as a pre-treatment to make glofitamab safer and more tolerable. Giving glofitamab with obinutuzumab pre-treatment may be safe, tolerable, and/or effective in treating patients with CNS lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety of glofitamab with obinutuzumab pre-treatment in patients with primary and secondary CNS lymphoma.

SECONDARY OBJECTIVES:

I. To estimate the overall response rate of glofitamab with obinutuzumab pre-treatment in primary and secondary CNS lymphoma.

II. To estimate the complete response rate, duration of response, duration of complete response, progression-free survival, event-free survival, and overall survival of glofitamab with obinutuzumab pre-treatment in primary and secondary CNS lymphoma.

EXPLORATORY OBJECTIVES:

I. To evaluate the degree to which glofitamab crosses the blood brain barrier (BBB) in CNS lymphoma and define biomarkers of response and toxicity to treatment.

II. To assess the utility of tocilizumab to address cytokine release syndrome in CNS lymphoma subjects treated with glofitamab.

III. To assess the utility of corticosteroids to address immune effector cell-associated neurotoxicity syndrome in CNS lymphoma subjects treated with glofitamab.

OUTLINE:

Patients receive obinutuzumab intravenously (IV) on day 1 of cycle 1 and glofitamab IV over 2-4 hours on days 8 and 15 of cycle 1 and on day 1 of subsequent cycles. Cycles repeat every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) or positron emission tomography (PET)/CT at screening and cerebrospinal fluid (CSF) and blood sample collection, brain magnetic resonance imaging (MRI) throughout the study. Patients with secondary CNS lymphoma also undergo CT or PET/CT throughout the study. Additionally, patients with baseline CSF involvement, may undergo lumbar puncture throughout the study.

After completion of study treatment, patients are followed up at 30 days and at 3, 6, 9, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Agreement to allow the use of archival tissue from diagnostic tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Age: ≥ 18 years
* Karnofsky performance status (KPS) ≥ 30
* Histologically confirmed primary or secondary CNS lymphoma. Tumor must be positive for CD20 by immunohistochemistry or flow cytometry on the most recent biopsy. Neuroimaging alone is acceptable in secondary CNS lymphoma cases where all of the following criteria are met: 1) brain MRI findings are consistent with CNS lymphoma, 2) the disease has been histologically documented in other sites, 3) the CNS lesions are concomitant with systemic progression, and 4) a brain biopsy would be unadvised per the treating provider.

  * Cohort 1: Primary CNS lymphoma
  * Cohort 2: Secondary CNS lymphoma
* Patients must not require urgent treatment initiation due to bulky or rapidly progressing CNS lymphoma that poses risk for impending critical brain failure. This includes > 5 mm of midline shift, radiographic evidence of impending brain herniation, or clinical evidence of significantly increased intracranial pressure such as papilledema
* Have failed methotrexate-based therapy or are ineligible/refuse high-dose methotrexate treatment (e.g. creatinine clearance [CrCl] < 50 mL/min, effusions, ascites etc)
* Measurable CNS lymphoma based on gadolinium enhancement of brain or spine MRI and/or positive CSF or intravitreal fluid cytology
* Fully recovered from the acute toxic effects (except alopecia) to ≤ grade 1 to prior anti-cancer therapy
* Alert and able to participate in a full neurological exam
* Without bone marrow involvement: Absolute neutrophil count (ANC) ≥ 1,000/mm^3

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement
* With bone marrow involvement: ANC ≥ 500/mm^3

  * NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement
* Without bone marrow involvement: Platelets ≥ 75,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment unless cytopenia is secondary to disease involvement
* With bone marrow involvement: Platelets ≥ 50,000/mm^3

  * NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment unless cytopenia is secondary to disease involvement
* Hemoglobin ≥ 8.0 g/dL
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (unless has Gilbert's disease, then ≤ 3.0 x ULN is allowed)
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN
* Alanine aminotransferase (ALT) ≤ 2.5 x ULN
* Creatinine clearance of ≥ 30 mL/min per 24 hour urine test or the Cockcroft-Gault formula
* If not receiving anticoagulants: International normalized ratio (INR) OR prothrombin (PT) ≤ 1.5 x ULN
* If on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants
* If not receiving anticoagulants: Activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN
* If on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants
* Seronegative for HIV antigen/antibody (Ag/Ab) combo

  * Individuals with a positive HIV test at screening are eligible provided, prior to enrollment, they are stable on antiretroviral therapy, have a CD4 count ≥ 200/uL, and have an undetectable viral load
* Seronegative for active hepatitis B virus (HBV) (surface antigen negative)

  * Participants with occult or prior hepatitis B infection (defined as positive total hepatitis B core antibody and negative hepatitis B virus surface antigen [HBsAg]) may be included if hepatitis B virus (HBV) deoxyribonucleic acid (DNA) is undetectable at the time of screening. Such participants must be willing to undergo HBV DNA testing on day 1 of every cycle and every 3 months for at least 12 months after the final cycle of study treatment and appropriate antiviral therapy as indicated
* Seronegative for HCV

  * Participants positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* Women of childbearing potential (WOCBP): Negative serum pregnancy test
* Agreement by females and males of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study and after completion of study treatment as described below separately for males and females

  * Female participants must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 18 months after pretreatment with obinutuzumab, 2 months after the final dose of glofitamab and 3 months after the final dose of tocilizumab (as applicable), whichever is longer. Women must refrain from donating eggs during this same period

    * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices
    * Hormonal contraceptive methods must be supplemented by a barrier method
  * For male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agree to refrain from donating sperm, as defined below:

    * With a female partner of childbearing potential or pregnant female partners, male participants must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 3 months after pretreatment with obinutuzumab, 2 months after the final dose of glofitamab or 2 months after the last dose of tocilizumab (as applicable), whichever is longer. Male participants must refrain from donating sperm during this same period
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the individual. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.
  * Childbearing potential defined as not being permanently surgically sterilized (men and women) or have not been free from menses for > 1 year (women only). Per this definition, a female participant with tubal ligation is considered to be of childbearing potential

Exclusion Criteria:

* Contraindication to any of the individual components of glofitamab or history of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies or known sensitivity or allergy to murine products
* Prior solid organ transplantation
* Prior treatment with systemic immunotherapeutic agents, including but not limited to, radio-immuno-conjugates, antibody-drug conjugates, immune/cytokines and monoclonal antibodies (mAbs) (e.g., anti cytotoxic T lymphocyte associated protein 4, anti PD-1, and anti PD-L1) within 2 weeks or five half-lives of the drug, whichever is shorter, prior to day 1 of protocol therapy
* Prior treatment with glofitamab or other CD20 x CD3 bispecific antibodies
* Prior use of systemic chemotherapy within 2 weeks of the start of cycle 1
* Prior treatment with intrathecal chemotherapy within 1 week of the start of cycle 1. Note, in patients with lymphoma restricted to the CSF and no other measurable sites of CNS disease, positive CSF cytology must be documented following the most recent administration of intrathecal chemotherapy
* Prior treatment with radiotherapy within 2 weeks prior to day 1 of protocol therapy

  * If patients have received radiotherapy within 4 weeks prior to day 1 of protocol therapy, patients must have at least one measurable lesion outside of the radiation field. Patients who have only one measurable lesion that was previously irradiated but subsequently progressed are eligible
* Prior treatment with chimeric antigen receptor T cell (CAR-T) therapy within 30 days prior to day 1 of protocol therapy
* Any investigational therapy for the purposes of treating cancer within 21 days prior to the start of cycle 1
* Corticosteroid use for purposes other than lymphoma symptom control

  * The use of inhaled corticosteroids is permitted
  * The use of mineralocorticoids for management of orthostatic hypotension is permitted.
  * The use of physiologic doses of corticosteroids for management of adrenal insufficiency is permitted.
  * Participants who require lymphoma symptom control during screening may receive steroids in the following manner:

    * Up to 50 mg/day of prednisone or equivalent may be used for lymphoma symptom control during screening
* History of other malignancy that could affect compliance with the protocol or interpretation of results:

  * Participants with a history of curatively treated basal or squamous cell carcinoma or melanoma of the skin or in situ carcinoma of the cervix at any time prior to the study are eligible
  * Participants with any malignancy appropriately treated with curative intent and the malignancy has been in remission without treatment for > 2 years prior to enrollment are eligible
  * Participants with low-grade, early-stage prostate cancer (Gleason score 6 or below, stage 1 or 2) with no requirement for therapy at any time prior to study are eligible
  * If the malignancy is expected to not require any treatment for at least 2 years (this exception should be discussed with the study PI)
* Unstable cardiac disease as defined by one of the following:

  * Cardiac events such as myocardial infarction (MI) within the past 3 months
  * NYHA (New York Heart Association) heart failure class III-IV
  * Unstable arrhythmias, or unstable angina
* Recent major surgery within 4 weeks prior to the start of cycle 1, other than for diagnosis
* Current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis or neurodegenerative disease with the exception of CNS lymphoma. Exceptions can be granted after discussion with the PI of the study

  * Participants with a history of stroke who have not experienced a stroke or transient ischemic attack in the past 2 years and have no residual neurological deficits, as judged by the investigator, are allowed
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
* History or presence of an abnormal electrocardiogram (ECG) that is clinically significant in the investigator's opinion
* Known or suspected active infection, or reactivation of a latent infection, whether bacterial, viral, fungal, mycobacterial, or other pathogens (excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics (for IV antibiotics this pertains to completion of last course of antibiotic treatment) within 4 weeks of dosing
* Active autoimmune disease requiring treatment with immune suppressive medications other than physiologic doses of steroids

  * Participants with a history of autoimmune-related hypothyroidism on a stable dose of thyroid-replacement hormone may be eligible
  * Participants with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
  * Participants with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only are eligible (e.g., participants with psoriatic arthritis are excluded) if all the following conditions are met:

    * Rash covers < 10% of body surface area
    * Disease is well controlled for the last 12 months and requires only low potency topical corticosteroids
* Clinically significant liver disease, including active viral or other hepatitis or cirrhosis
* Live, attenuated vaccine within 4 weeks before study treatment infusion on day 1 of cycle 1 or anticipation that such a live, attenuated vaccine will be required during the study. Live vaccines during the study and until participants B cells recover, are prohibited

  * Influenza vaccination should be given during influenza season only. Participants must not receive live, attenuated influenza vaccine at any time during the study treatment period
* Suspected active or latent tuberculosis (as confirmed by a positive interferon gamma release assay)
* Participants with a history of progressive multifocal leukoencephalopathy
* Females only: Pregnant or breastfeeding or intention of becoming pregnant during the study or within 18 months after pretreatment with obinutuzumab or 2 months after the final dose of glofitamab, whichever is longer
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2029-01-02 (Estimated); Study Completion 2029-01-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 or higher non-hematologic toxicity that does not resolve to grade 1 or better within 7 days | During first 2 cycles of treatment (cycle length = 21 days)
  For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided. For categorical variables, counts and percentages will be provided. Observed toxicities will be summarized by type, severity, and attribution.
Incidence of grade 3 or 4 thrombocytopenia associated with grade >= 3 bleeding | During first 2 cycles of treatment (cycle length = 21 days)
  For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided. For categorical variables, counts and percentages will be provided. Observed toxicities will be summarized by type, severity, and attribution.
Incidence of grade 4 neutropenia or grade 4 thrombocytopenia (without clinically significant bleeding) that lasts > 14 days | During first 2 cycles of treatment (cycle length = 21 days)
  For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided. For categorical variables, counts and percentages will be provided. Observed toxicities will be summarized by type, severity, and attribution.
Incidence of grade >= 3 cytokine release syndrome (CRS) not resolving to grade 1 or better within 7 days | During first 2 cycles of treatment (cycle length = 21 days)
  For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided. For categorical variables, counts and percentages will be provided. Observed toxicities will be summarized by type, severity, and attribution.
Incidence of grade 4 CRS | During first 2 cycles of treatment (cycle length = 21 days)
  For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided. For categorical variables, counts and percentages will be provided. Observed toxicities will be summarized by type, severity, and attribution.
Incidence of any emergent grade 3 neurologic toxicity | During first 2 cycles of treatment (cycle length = 21 days)
  For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided. For categorical variables, counts and percentages will be provided. Observed toxicities will be summarized by type, severity, and attribution.
Incidence of emergent grade 4 neurologic toxicity | During first 2 cycles of treatment (cycle length = 21 days)
  For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided. For categorical variables, counts and percentages will be provided. Observed toxicities will be summarized by type, severity, and attribution.
Incidence of any grade 5 toxicity | During first 2 cycles of treatment (cycle length = 21 days)
  For continuous variables, descriptive statistics such as number, mean, standard deviation, standard error, median (range) etc. will be provided. For categorical variables, counts and percentages will be provided. Observed toxicities will be summarized by type, severity, and attribution.

SECONDARY OUTCOMES:
Overall response rate (ORR) | From start of protocol therapy to disease progression and/or start of other anti-lymphoma therapy, assessed up to 24 months
  Will be defined as achieving a best response of complete response (CR) or partial response (PR). Will be tabulated by the response categories. ORR will be estimated as a percentage along with the 95% exact binomial confidence interval.
CR rate | From start of protocol therapy to disease progression and/or start of other anti-lymphoma therapy, assessed up to 24 months
  Will be tabulated by the response categories. CR rate will be estimated as a percentage along with the 95% exact binomial confidence interval.
Duration of response (DOR) | From first achievement of PR or CR to time of progression, relapse, or death, whichever is earlier, assessed up to 24 months
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median DOR will be estimated when available.
Duration of CR (DOCR) | From first achievement of CR to time of progression, relapse or death, whichever is earlier, assessed up to 24 months
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median DOCR will be estimated when available.
Progression-free survival (PFS) | From start of protocol treatment to time of progression, relapse, or death due to any cause, whichever occurs earlier, assessed up to 24 months
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median PFS will be estimated when available.
Event-free survival (EFS) | From the start of protocol treatment to time of progression, relapse, start of any new anti-lymphoma therapy, or death due to any cause, whichever occurs earlier, assessed up to 24 months
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median EFS will be estimated when available.
Overall survival (OS) | From start of protocol treatment to time of death due to any cause, assessed up to 24 months
  Will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error; 95% confidence interval will be constructed based on log-log transformation. Median OS will be estimated when available.

CONTACTS AND LOCATIONS:
Overall Officials: James Godfrey, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States